CLINICAL TRIAL: NCT02801500
Title: Superior Bilioenteric Anastomosis by Magnetic Compressive Technique: A Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Superior Bilioenteric Anastomosis by Magnetic Compressive Technique
Acronym: CTREG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Shaanxi Provincial People's Hospital (Other); Tang-Du Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2015-001
Record Dates: First submitted 2016-05-29; First posted 2016-06-16 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Hilar Cholangiocarcinoma; Bile Duct Injury; Choledochal Cyst; Biliary Calculi
Keywords: bilioenteric anastomosis
MeSH Terms: conditions — Klatskin Tumor; Choledochal Cyst; Gallstones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic Compressive Anastomosis (Experimental): A magnetic device will be used during bilioenteric anastomosis.
  Interventions: Device: Magnetic Compressive Anastomosis
- Traditional Manual Anastomosis (Active Comparator): A handsewn technique will be used during bilioenteric anastomosis.
  Interventions: Procedure: Manual Anastomosis

INTERVENTIONS:
Device: Magnetic Compressive Anastomosis — The magnetic compressive anastomosis device will be used to complete the anastomosis during bilioenteric anastomosis.
  Arms: Magnetic Compressive Anastomosis
Procedure: Manual Anastomosis — A handsewn technique will be used to complete the anastomosis during bilioenteric anastomosis.
  Arms: Traditional Manual Anastomosis

SUMMARY:
The purpose of this study is to determine whether the magnetic compressive anastomosis has a better outcomes than traditional manual anastomosis on superior bilioenteric anastomosis.

DETAILED DESCRIPTION:
The superior bilioenteric anastomosis is one of the most common and difficult operations in Hepatobiliary Surgery. The traditional manual anastomosis has become one of the main prognosis factors because of the length of suture time, the difficulty of operation, the high incidence of anastomotic leakage and stricture. Magnetic compressive anastomosis can realize the fast anastomosis, reduce the difficulty, and reduce the incidence of anastomotic leakage and stricture. Currently, the majority of studies of magnetic compressive bilioenteric anastomosis are merely confined within clinical case report and single-center, small sample, retrospective study, thus they are lack of convictive evidence of evidence-based medicine for the security, reliability and convince.

This study is a multicenter, prospective, randomized controlled trial. To evaluate the security, reliability and convince of magnetic compressive superior bilioenteric anastomosis, this study compared the incidence of anastomotic leakage and stricture between magnetic compressive anastomosis and traditional manual anastomosis among patients who need superior bilioenteric anastomosis operation. The study design plan to enroll 70 patients and divide into Study Group (Group A: Magnetic compressive anastomosis) and Control Group (Group B: traditional manual anastomosis) as 1:1 ratio randomly by stratification factors. The incidence of anastomotic leakage and stricture, length of bilioenteric anastomosis time, value of serum bilirubin, length of discharge time of magnetic device and mean time of hospital stay will be evaluated. The patients will drop out of the study if adverse events happen, active request for dropping out, new-onset severe disease or death. The primary and secondary end point will be observed by regular follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 to 75
* Patients' gender was not limited
* Patients who were well-diagnosed and had the indication for superior bilioenteric anastomosis.
* Patients whose lifetimes will be longer than 12 months.
* Patients who are willing to join this clinical trial and informed consent form voluntarily.

Exclusion Criteria:

* Woman during pregnancy or lactation or anyone with mental disorder
* The wall of hepatic duct or jejunum was too thick so that the attractive force of magnetic device cannot meet the requirements of compression.
* Any anatomical variation in bile ducts system or the inner diameter is too small so that the magnetic device cannot place in.
* Any foreign body has been implanted in body, such as heart pacemaker.
* Surgical contraindication, including:

Child-Pugh C with hepatic encephalopathy Anyone with heart, lung, kidney dysfunction or other organ dysfunction, and cannot tolerate surgery.Hepatic ducts stone disease, who was diagnosed as Acute Cholangitis of Severe Type, especially complicated with bacteremia or septic shock. End stage disease, complicated with biliary cirrhosis or portal hypertension.Patients with long-term obstructive jaundice, dehydration, electrolyte disturbance or coagulation defects; Patients have the tendency or history of bleeding.

* Any other disease in perioperation periods which needs MRI examination in the next 8 weeks post operation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Bilioenteric anastomotic leakage | 1 month post operation

SECONDARY OUTCOMES:
Length of bilioenteric anastomosis time | during operation
Number of patients who have discharged the device on the date expected. | 1 to 4 weeks postoperation
Number of patients who have been diagnosed as discharge disorder of magnetic device | less than 1 week or more than 4 weeks
average length of postoperative hospital stay | 3 months
Times of pathological examination of bile duct's remnant of Klatskin' tumor | during operation
Bilioenteric anastomotic stricture | Time Frame: 1,3,6,12-month post operation

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sicklick JK, Camp MS, Lillemoe KD, Melton GB, Yeo CJ, Campbell KA, Talamini MA, Pitt HA, Coleman J, Sauter PA, Cameron JL. Surgical management of bile duct injuries sustained during laparoscopic cholecystectomy: perioperative results in 200 patients. Ann Surg. 2005 May;241(5):786-92; discussion 793-5. doi: 10.1097/01.sla.0000161029.27410.71. PMID 15849514
- [Result] House MG, Cameron JL, Schulick RD, Campbell KA, Sauter PK, Coleman J, Lillemoe KD, Yeo CJ. Incidence and outcome of biliary strictures after pancreaticoduodenectomy. Ann Surg. 2006 May;243(5):571-6; discussion 576-8. doi: 10.1097/01.sla.0000216285.07069.fc. PMID 16632990
- [Result] Frattaroli FM, Reggio D, Guadalaxara A, Illomei G, Pappalardo G. Benign biliary strictures: a review of 21 years of experience. J Am Coll Surg. 1996 Nov;183(5):506-13. PMID 8912621
- [Result] Yan JQ, Peng CH, Ding JZ, Yang WP, Zhou GW, Chen YJ, Tao ZY, Li HW. Surgical management in biliary restricture after Roux-en-Y hepaticojejunostomy for bile duct injury. World J Gastroenterol. 2007 Dec 28;13(48):6598-602. doi: 10.3748/wjg.v13.i48.6598. PMID 18161934
- [Result] Avaliani M, Chigogidze N, Nechipai A, Dolgushin B. Magnetic compression biliary-enteric anastomosis for palliation of obstructive jaundice: initial clinical results. J Vasc Interv Radiol. 2009 May;20(5):614-23. doi: 10.1016/j.jvir.2009.01.019. PMID 19393505
- [Result] Chopita N, Vaillaverde A, Cope C, Bernedo A, Martinez H, Landoni N, Jmelnitzky A, Burgos H. Endoscopic gastroenteric anastomosis using magnets. Endoscopy. 2005 Apr;37(4):313-7. doi: 10.1055/s-2005-861358. PMID 15824939
- [Result] Stepanov EA, Vasil'ev GS, Nikolaev VV. [The treatment of intestinal fistulae in children by applying a by-pass anastomosis using magnetic devices]. Khirurgiia (Mosk). 1992 Nov-Dec;(11-12):93-5. Russian. PMID 1294807
- [Result] Fan C, Ma J, Zhang HK, Gao R, Li JH, Yu L, Wu Z, Lv Y. Sutureless intestinal anastomosis with a novel device of magnetic compression anastomosis. Chin Med Sci J. 2011 Sep;26(3):182-9. doi: 10.1016/s1001-9294(11)60046-1. PMID 22207929